CLINICAL TRIAL: NCT02500238
Title: Comparison of Smoking and Vaping in Families
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500475; OCR14742 (Other: University of Florida)
Record Dates: First submitted 2015-07-08; First posted 2015-07-16 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva, urine, and toenail clippings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: This group will provide 2 breath carbon monoxide (reading of ≤ 6 parts per million) and a saliva sample, urine sample, and toe nail clippings will be taken from this group.
  Interventions: Other: Saliva sample; Other: Urine Sample; Other: Toe nail clippings; Other: Breath carbon monoxide test
- Smoking: This group will provide 1 breath carbon monoxide test (reading of ≤ 6 parts per million) and a saliva sample, urine sample, and toe nail clippings.
  Interventions: Other: Saliva sample; Other: Urine Sample; Other: Toe nail clippings; Other: Breath carbon monoxide test
- Vaping: This group will provide 2 breath carbon monoxide test (reading of ≤ 6 parts per million) and a saliva sample, urine sample, and toe nail clippings.
  Interventions: Other: Saliva sample; Other: Urine Sample; Other: Toe nail clippings; Other: Breath carbon monoxide test

INTERVENTIONS:
Other: Saliva sample — All participants will provide a saliva sample.
Other: Urine Sample — All participants will provide a urine sample.
Other: Toe nail clippings — All participants will provide toe nail clippings.
Other: Breath carbon monoxide test — All participants will provide breath carbon monoxide tests

SUMMARY:
Electronic cigarette use may be less harmful than cigarettes in adults, however, limited data exists examining passive electronic cigarette exposure and child health outcomes. The current study seeks to compare health-related outcomes among youth who reside with non-smokers, cigarette smokers, and electronic cigarette users. The investigators propose to conduct a small pilot study with 30 youth, ages 6-17 and a caregiver. Three groups of 10 parent-child dyads will be recruited: 1) control group: parents who are non-smokers/non-vapers, 2) smoking group: parents who are exclusive cigarette smokers, and 3) vaping group: parents who are exclusively ECIG users. Groups will be compared across the following variables: child lung function and biomarkers of nicotine.

DETAILED DESCRIPTION:
The current study seeks to compare health-related outcomes among youth who reside with non-smokers, cigarette smokers, and electronic cigarette users.

Control Group: will consist of participants ages 6 - 17 who live in a home with adults who do not smoke. A brief breathing test will verify a non-smoker and/or are not around a certain amount of smoke in the environment (live with a smoker). The participant will be asked to complete a series of brief questionnaires that asks about basic demographic information, medical history, and that asks about their smoking history. The participant's will also be asked to complete two 5 minute breathing tests, provide a sample of saliva, a urine sample, and have their toe nails clipped.

Vaping Group: will consist of participants ages 6 -17 who live in a home with adults who currently use electronic cigarettes. A brief breathing test will verify a non-tobacco smoker and/or are not around a certain amount of smoke in the environment (live with a tobacco smoker). The participant will be asked to complete a series of brief questionnaires that asks about basic demographic information, smoking or vaping history and patterns of use, and medical history. The participant will be asked to complete two 5 minute breathing tests, provide a sample of saliva, a urine sample, and have their toe nails clipped.

Smoking Group: will consist of participants ages 6 - 17 who live in a home with adults who currently smoke cigarettes. Participants will then be asked to complete a series of brief questionnaires that asks about basic demographic information, smoking or vaping history and patterns of use, and medical history. The participant will also be asked to complete two 5 minute breathing tests, provide a sample of saliva, a urine sample, and have their toe nails clipped.

ELIGIBILITY:
Inclusion Criteria:

For the control group the caregiver must self-report:

1. never smoking or not smoking for at least the past 12 months;
2. that no one living in the home is a current smoker or has smoked in the home for the past 6 months; and
3. have a breath carbon monoxide reading of ≤ 6ppm.

For the smoking group caregivers must:

1. smoke at least 10 cigarettes per day for the past year;
2. indicate that they smoke in the car or home ≥ 3 times per week; and
3. do not use non-cigarette tobacco (e.g., cigars, chewing tobacco).

For the vaping group caregivers must:

1. exclusively use EC for the past 3 months (no cigarette or other tobacco use); and
2. no one living in the home is a current tobacco smoker or has smoked in the home for the past 6 months; and
3. have a breath carbon monoxide reading of ≤ 6ppm.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In order to be included in the study, parents must: 1) be a legal guardian of a child between the ages of 6-17 (if caregiver has more > 1 child between 6-17 years; 2) be aged 18-65 years; and 3) be fluent in English. Additionally, the child must reside in the same home as the caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Assessment of lung function | Day 1
  Child lung function will be measured at the study visit. Forced expiratory volume in the first second will be assessed.

SECONDARY OUTCOMES:
Assessment of cotinine in saliva | Day 1
  Child saliva samples will be collected at the study visit. Samples will be assessed for cotinine levels.
Assessment of cotinine in urine | Day 1
  Child urine samples will be collected at the study visit. Samples will be assessed for cotinine levels.
Assessment of nicotine in toenail clippings | Day 1
  Child toenail samples will collected at the study visit. Samples will be assessed for nicotine levels.
Assessment of cotinine in toenail clippings | Day 1
  Child toenail samples will be collected at the study visit. Samples will be assessed for cotinine levels.
Assessment of tobacco specific nitrosamine in toenail clippings | Day 1
  Child toenail samples will be collected at the study visit. Samples will be assessed for NNAL levels.
Assessment of tobacco specific nitrosamine in urine | Day 1
  Child urine samples will be collected at the study visit. Samples will be assessed for NNAL levels.

CONTACTS AND LOCATIONS:
Overall Officials: David A Fedele, Ph.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Uf Ctsi Crc, Gainesville, Florida
  - OUHSC, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided